CLINICAL TRIAL: NCT04437316
Title: Effect of Low Level Laser Therapy After Wisdom Tooth Removal on Swelling, Pain and Mouth Opening in a Randomized, Double-blind Split-mouth Study
Brief Title: Effect of Low Level Laser Therapy After Wisdom Tooth Removal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-00949
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Tooth, Impacted; Wound Heal; Quality of Life
Keywords: Wisdom tooth; Low Level Laser
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Intervention Model Description: split-mouth design
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Level Laser (Active Comparator): therapeutic laser
  Interventions: Device: Use of Low level Laser after wisdom tooth removal
- Placebo Low Level Laser (Placebo Comparator): non-therapeutic laser
  Interventions: Device: Use of Low level Laser after wisdom tooth removal

INTERVENTIONS:
Device: Use of Low level Laser after wisdom tooth removal — Directly after the wisdom teeth removal of the right/left side, one of the low level laser (therapeutic and non-therapeutic (Placebo)) is used.

SUMMARY:
The aim is to test the effect of low level laser therapy on the relief of symptoms after wisdom tooth removal.

DETAILED DESCRIPTION:
Each Patient will get all four wisdom teeth removed, left and right side separately. After the operation, low level laser therapy is applied intra- and extraorally. Two different lasers are used, one for each side. The two lasers look identical. Only one of the lasers has therapeutic light, the other one shows just non-therapeutic red light. The effect of the low level laser is measured by several parameters and they are compared with the other side. These parameters are pain, swelling and mouth opening. The selection of the lasers to the sides is double-blind and randomized.

ELIGIBILITY:
Inclusion Criteria:

* Indication for prophylactical wisdom tooth removal
* 4 wisdom teeth

Exclusion Criteria:

* pregnancy
* taking blood thinners
* known infectious diseases
* untreated diabetes mellitus
* taking immunosuppressants
* Previous infections in the area of the wisdom teeth
* smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 3 days after wisdom tooth removal
  Measurement of Pain with a visual analogue scale (VAS) 0-10

SECONDARY OUTCOMES:
Postoperative Pain | 7 days after wisdom tooth removal
  Measurement of Pain with a visual analogue scale (VAS) 0-10
Postoperative Swelling | 3 and 7 days after wisdom tooth removal
  Measurement of swelling with an extraoral scan
Postoperative Mouth opening | 3 and 7 days after wisdom tooth removal
  Measurement of mouth opening

CONTACTS AND LOCATIONS:
Overall Officials: Martin Ruecker, Prof., Study Director — Clinic for maxillofacial and oral surgery
Locations (1):
- Center of dental medicine, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No